CLINICAL TRIAL: NCT05432830
Title: Sex Differences in E-Cigarette Flavor Sensory Perception As It Relates to Appeal and Reinforcing Efficacy Among Adult Smokers: Study 1
Brief Title: Sex Differences in E-cig Perception: Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000032981; 1K01DA056494-01 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Nicotine Addiction; E-Cig Use; Cigarette Smoking; Sex Differences
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Within subject design, all participants will receive all flavors
Who Masked: Participant, Investigator
Masking Description: Double blind, both participant and investigator will be blind to e-liquid being administered
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental E-Liquid Order "A" (Experimental): All participants will be given all e-liquids (i.e. 3 flavor conditions all containing nicotine) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across 3 visits).
  Interventions: Other: E-liquid Flavor 1; Other: E-liquid Flavor 2; Other: E-liquid Flavor 3
- Experimental E-Liquid Order "B" (Experimental): All participants will be given all e-liquids (i.e. 3 flavor conditions all containing nicotine) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across 3 visits).
  Interventions: Other: E-liquid Flavor 1; Other: E-liquid Flavor 2; Other: E-liquid Flavor 3
- Experimental E-Liquid Order "C" (Experimental): All participants will be given all e-liquids (i.e. 3 flavor conditions all containing nicotine) in this within subject cross-over design study. Participants will be randomized in the order in which they receive the flavor conditions (across 3 visits).
  Interventions: Other: E-liquid Flavor 1; Other: E-liquid Flavor 2; Other: E-liquid Flavor 3

INTERVENTIONS:
Other: E-liquid Flavor 1 — E-liquid containing 36mg/ml pronated nicotine will be administered with sweet e-cigarette flavor.
Other: E-liquid Flavor 2 — E-liquid containing 36mg/ml pronated nicotine will be administered with cooling e-cigarette flavor.
Other: E-liquid Flavor 3 — E-liquid containing 36mg/ml pronated nicotine will be administered with unflavored e-cigarette flavor.

SUMMARY:
The primary objective is to examine the influence of sex on sensory effects, appeal, and reinforcing value of nicotine containing e-cigs in popular flavor components; sweet and cooling.

DETAILED DESCRIPTION:
This study looks at the effect of sex on the sensory effects of flavor components in e-cigarettes. Regular combustible tobacco users will sample 3 different flavored e-cigarettes containing nicotine in a human lab paradigm.

ELIGIBILITY:
Inclusion Criteria:

* 21-44 years old
* Able to read/write
* Current cigarette smoking
* Recent E-cig Exposure (>/= 10 uses in past 6 mo.)
* Urine cot >200ng/ml
* Willing to abstain from nicotine/tobacco 6-8hrs prior to lab session
* Not looking to quit

Exclusion Criteria:

* Untreated chronic medical conditions
* Non-stable Rx medication
* Illicit drug use
* Pregnant, trying to become pregnant, breastfeeding
* Not fully vaccinated for Coronavirus (e.g. COVID-19)

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Appeal | immediately after intervention, up to 15 minutes
  Change in appeal at each flavor as measured by the computerized Labeled Hedonic Scale (LHS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Labeled Hedonic Scale (LHS) is a bipolar category ratio scale that ranges from -100 (most disliked) to 100 (most liked), with 'neither liked nor disliked' as midpoint.
Sensory Effects | immediately after intervention, up to 15 minutes
  Change in sweetness, coolness, irritation, and bitterness at each flavor as measured by the computerized Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Reinforcing Efficacy | immediately after intervention, up to 15 minutes
  Change in reinforcing value at each flavor. Participants will use the multiple choice procedure to self-report their responses using a computer mouse to indicate where on the scale response falls. Following each puffing bout, participants will be asked to make discrete hypothetical choices between 10-puffs of the e-cig they had just used or a series of 44 monetary values ($0.25-$15.06). The minimum monetary value at which money is chosen over the e-cig puffs is a contingency-based estimate of e-cig value. At the end of each lab session, participants will be given a choice between another 10 e-cig puffs or one of the monetary amounts they picked in the Multiple Choice Procedures completed earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Davis, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT05432830/ICF_000.pdf